CLINICAL TRIAL: NCT00900601
Title: Surgical Treatment of Pelvic Joint Instability in Patients With Severe Pelvic Girdle Pain After Pregnancy and Trauma - A Study to Measure Effect of Surgery, Analysis of Clinical Tests and Detection of Sacroiliac Instability Using RSA.
Brief Title: Surgical Treatment of Pelvic Joint Instability in Patients With Severe Pelvic Girdle Pain After Pregnancy and Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other)
Responsible Party: Principal Investigator, Thomas Johan Kibsgård, Consultant, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UUS nr: 28125409; REK: 1.2006.1574
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2017-09

CONDITIONS: Pelvic Joint Instability; Pelvic Pain
Keywords: Sacroiliac pain; Sacroiliac instability; Pelvic girdle pain; Sacroiliac arthrodesis; Arthrodesis; Surgery
MeSH Terms: conditions — Pelvic Pain; Pelvic Girdle Pain; Ankylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sacroilliac fusion (Experimental): Pastient are treated with sacroiliac joint arthrodesis to the sacroiliac joint and symphysis
  Interventions: Procedure: Arthrodesis to the sacroiliac joint and symphysis

INTERVENTIONS:
Procedure: Arthrodesis to the sacroiliac joint and symphysis — Standard surgical procedures will be used. When the patient has isolated pain in the symphysis isolated fixation will be performed. A 2x2 cm large bone block will be removed and replaced with spongy bone. For fixation the Matta-plate will be applied.
  To the sacroiliac joint we use an anterior approach. A 2x1,5 cm large bone block will be removed and replaced with spongy bone from the iliac crest. For joint fixation we either use 2 plates or sacroiliac screws. The same procedure will be used on the other side in the cases with bilateral symptoms. Only one side will be operated at a time. After one year it will be decided if it's necessary to perform contralateral surgery.

SUMMARY:
Pelvic girdle pain (PGP) related to pregnancy is a common reason to sick leave during pregnancy. Low back pain and PGP affects about 50% of women during pregnancy. Most of the women recover, however about 10% of the women still have complaints after birth. Most patients have positive effect from conservative treatment, but unfortunately some do still have much pain despite intensive conservative rehabilitation. Surgery has been tried on these women with various results. Surgical treatment is controversial and there is a lack of documentation. The investigators will operate 20 patients with arthrodesis to the sacroiliac joint and symphysis. Radiostereometric analysis (RSA) will be used to evaluate the joint movement in different part of the process.

Hypothesis: Severe pelvic girdle pain is caused by pelvic joint instability in some cases and surgically fixation of the affected joints can help these women to get back to a normal life.

ELIGIBILITY:
Inclusion Criteria:

* Pain in one or more pelvic joints.
* Minimum 2 positive clinical tests.
* High pain and disability score
* Tried adequate physiotherapy without effect.

Exclusion Criteria:

* Known psychiatric diagnosis
* Other spine pathology
* CT verified ankylosis
* BMI>30

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Kibsgaard, PhD student, Principal Investigator — Oslo university hosptal - Ullevaal
Locations (1):
- Oslo university hospital - Ulllevaal, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study period, from 2007 and 2010, a total of 20 patients with PGP were referred Oslo University Hospital, but only 9 patients met the study's inclusion criteria.
Groups:
- Sacroliac Joint Fusion: Patients treated with sacroiliac joint fusion
Period: Overall Study
Arm/Group | Sacroliac Joint Fusion
Started | 9
Completed | 8
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sacroliac Joint Fusion
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 40 [33 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Norway | 9
Duration of pain [Median (Full Range); unit: years] | 11 [2 to 25]
BMI [Median (Full Range); unit: kg/m2] | 25 [20 to 30]
Etiology [Count of Participants; unit: Participants]
  Post preganancy | 7
  Trauma | 2
Unilateral/Bilateral [Count of Participants; unit: Participants]
  Unilateral pain | 1
  Bilateral pain | 8

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index (ODI)
Description: Oswestry Disability Index is a 10 item questionnaire comprises 10 questions about physical function. Each item has a 0-5 scale and the raw score is multiplied by 2 and the sum is the total score. Zero represents excellent physical function and 100 is more or less bedridden. This is the most used outcome measure in low back pain studies.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sacroliac Joint Fusion
Number analyzed (Participants) | 8
units on a scale
  Baseline | 54 [48 to 60]
  One year | 37 [34 to 40]

2. Primary Outcome: Visual Analogue Scale (VAS) 0 to 10
Description: Visual Analogue Scale is a 0 -10 scale. Zero is no pain and 10 is the worst pain you can imagine. In this study the patients were asked to report the morgning and evening pain by this scale.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sacroliac Joint Fusion
Number analyzed (Participants) | 8
units on a scale
  Baseline | 81 [76 to 87]
  One year | 57 [49 to 61]

3. Secondary Outcome: Healing Measured by CT
Description: Number of participants with healing as measured by CT data. The outcome was radiological healing vs no signs of radiological healing. In order to be classified as healed the CT scans had to show Clear signs of bone bridging across the sacroiliac joint.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sacroliac Joint Fusion
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sacroliac Joint Fusion
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sacroliac Joint Fusion (N=8)
Nerve damage (Nervous system disorders) | 1 (1) — Nervedamage to the lumbosacral plexus
Infection (Infections and infestations) | 1 (1) — Deep wound infection
Loss of bladder sensation (Nervous system disorders) | 1 (1) — Loss of bladder sensation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sacroliac Joint Fusion (N=8)
Transient sensitivity loss to the lateral femoral cutaneous nerve (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No